CLINICAL TRIAL: NCT03603665
Title: A Phase I, Double-Blind, Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of NTM-1633 vs Placebo Administered Intravenously in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of NTM-1633 vs Placebo Administered Intravenously in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0023; HHSN272201300017I
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2018-07-17

CONDITIONS: Botulism
Keywords: Botulism; Dose Escalation; Double-Blind; NTM-1633; Pharmacokinetics; Phase I; Safety
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Experimental): Single intravenous (IV) infusion of 0.033 mg/kg NTM-1633 (N=6) or matching Placebo (N=2) using an infusion pump over 60 minutes
  Interventions: Biological: NTM-1633; Other: Placebo
- Arm B (Experimental): Single IV infusion of 0.165 mg/kg NTM-1633 (N=6) or matching Placebo (N=2) using an infusion pump over 60 minutes
  Interventions: Biological: NTM-1633; Other: Placebo
- Arm C (Experimental): Single IV infusion of 0.330 mg/kg NTM-1633 (N=6) or matching Placebo (N=2) using an infusion pump over 60 minutes
  Interventions: Biological: NTM-1633; Other: Placebo

INTERVENTIONS:
Biological: NTM-1633 — NTM-1633 is an equimolar mixture of three IgG1 monoclonal antibodies (mAb), referred to as XE02, XE06, and XE17 which bind to non-overlapping epitopes on Botulinum Neurotoxin (BoNT/E). Administered as a single intravenous infusion of NTM-1633 over one hour.
Other: Placebo — 0.9% Sodium Chloride Injection administered as a single intravenous infusion over one hour.

SUMMARY:
This is a Phase I, single-center, double-blind, placebo-controlled dose escalation trial of three dose cohorts (A: 0.033 mg/kg, B: 0.165 mg/kg, and C: 0.33 mg/kg). The purpose of this study is to evaluate the safety and tolerability of NTM-1633 in healthy adults. This is a first-in-human study consisting of three cohorts of eight subjects each. Dosing for each cohort is as follows: Two sentinel subjects will be administered a single 1-hour infusion (one NTM-1633, one placebo). No more than two subjects per day thereafter (at least 24 hrs will elapse between the dosing of each two subjects) will be dosed in the same manner until all subjects are dosed. Dose escalation will not occur until safety data through Day 8 is reviewed by the Safety Review Committee (SRC). Objective dose-escalation criteria and safety evaluations will be utilized. The study duration will be for approximately 8 months. Subjects in Cohort A will participate for approximately 17 weeks and Subjects in Cohorts B and C will participate approximately 21 weeks. Primary Objective: To assess the safety and tolerability of escalating doses of NTM-1633 administered intravenously in healthy adults.

DETAILED DESCRIPTION:
This is a Phase I, single-center, double-blind, placebo-controlled dose escalation trial of three dose cohorts (A: 0.033 mg/kg, B: 0.165 mg/kg, and C: 0.33 mg/kg). The purpose of this study is to evaluate the safety and tolerability of NTM-1633 in healthy adults. This is a first-in-human study consisting of three cohorts of eight subjects each. Dosing for each cohort is as follows: Two sentinel subjects will be administered a single 1-hour infusion (one NTM-1633, one placebo). No more than two subjects per day thereafter (at least 24 hrs will elapse between the dosing of each two subjects) will be dosed in the same manner until all subjects are dosed. Dose escalation will not occur until safety data through Day 8 is reviewed by the Safety Review Committee (SRC). Objective dose-escalation criteria and safety evaluations will be utilized. The study duration will be for approximately 8 months. Subjects in Cohort A will participate for approximately 17 weeks and Subjects in Cohorts B and C will participate approximately 21 weeks. Primary Objective: To assess the safety and tolerability of escalating doses of NTM-1633 administered intravenously in healthy adults. Secondary Objectives: 1) To assess the pharmacokinetic characteristics of NTM-1633 following a single intravenous administration; 2) To assess the immunogenicity of NTM-1633 following a single intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood and signed.
2. Healthy male or healthy, non-pregnant, non-lactating female.
3. Willingness to comply and be available for all protocol procedures including inpatient confinement for 36 - 48 hours.
4. Age between 18 and 45 years, inclusive on the day of infusion.
5. Body Mass Index (BMI) of > / =18.5 and < 35 kg/m^2.
6. If the subject is female and of childbearing potential, she has a negative serum pregnancy test at screening and negative urine test within 24 hours prior to infusion.

   * A woman is considered of childbearing potential unless post-menopausal (> / = 1 year without menses) or surgically sterilized via bilateral oophorectomy, or hysterectomy or bilateral tubal ligation or successful Essure placement with documented confirmation test at least 3 months after the procedure.
7. If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use acceptable contraception up to visit 12 of the study.

   * Acceptable contraception methods are restricted to effective devices (Intrauterine Contraceptive Devices, NuvaRing(R)) or licensed hormonal products with use of method for a minimum of 28 days prior to dosing, condoms or diaphragm with spermicidal agents, monogamous relationship with a vasectomized partner
8. The hemoglobin, platelet count, white blood cell count and absolute neutrophil count are within normal limits at the screening visit.
9. The urine dipstick results on protein, glucose and blood are negative or trace.

   * Menstruating females failing inclusion criteria due to a positive blood on urine dipstick may be retested following cessation of menses.
10. Chemistry screening laboratory tests are in the normal reference range.

    * The following exceptions to laboratory normal reference ranges are allowed: Creatinine, Blood Urea Nitrogen (BUN), total bilirubin, AST, ALT, lipase, amylase, Prothrombin Time (PT), Partial Thromboplastin Time (PTT) below the lower limit of normal (LLN); CK less than 400mg/ml; Glucose, potassium, total protein, and alkaline phosphatase with a toxicity grade of 1 is allowable; albumin above the upper limit of normal (ULN).

      * Laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to laboratory error may be repeated once.
      * Abnormalities in mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV), and nucleated red blood cell count (NRBC CT), which are included in a complete blood count with differential, will not be exclusionary.
11. Has adequate venous access for the infusion.
12. The urine drug screen is negative.
13. Breathalyzer test is negative.
14. Available for follow-up for the duration of the study.
15. Agrees not to participate in vigorous activity 72 hours prior to dosing through day 15 post dosing.

Exclusion Criteria:

1. History of a chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject.

   * Chronic medical conditions include diabetes; Asthma requiring use of medication in the year before screening; Autoimmune disorder such as lupus, Wegener's, rheumatoid arthritis, thyroid disease; Coronary artery disease; Chronic hypertension; History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease (except previous asthma which has required no treatment for the past year)
2. History of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins.

   * Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema
3. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 450 milliseconds)
4. Clinically significant abnormal electrocardiogram at screening.

   * Clinically significant abnormal ECG results include: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator
5. Positive serology results for HIV, HBsAg, or HCV antibodies
6. Febrile illness with temperature > 37.6 degrees Celsius within 7 days of dosing
7. Pregnant or breastfeeding
8. Donated blood within 56 days of enrollment (day -1)
9. Known allergic reactions to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure
10. Treatment with another investigational drug within 28 days of dosing
11. Treatment with a monoclonal antibody at any time in the past
12. Receipt of antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
14. Use of H1 antihistamines or beta-blockers within 5 days of dosing
15. Use of any prohibited medication within 28 days prior to study entry or planned use during the study period

    * Prohibited medications include immunosuppressives (except Nonsteroidal Anti-Inflammatory Drugs [NSAIDS]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents; any vaccine (licensed or investigational). If study activities overlap with the influenza season, subjects will be instructed to delay influenza vaccination until after Day 57 (Visit 11)
16. Previous exposure to botulinum toxin, receipt of antibodies against botulinum toxin, or previous treatment with equine antitoxin
17. Any previous injection or planned injection within 4 months after enrollment of botulinum toxin for cosmetic reasons, spastic dysphonia, torticollis, or any other reason
18. Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety
19. Plans to enroll or is already enrolled in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period

    * Includes trials that have a study intervention such as a drug, biologic, or device
20. Is a study site employee or staff who are paid entirely or partially by the OCRR contract for the DMID-funded trial

    * Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators
21. Systolic blood pressure >140 mm Hg or diastolic blood pressure > 90 mm Hg
22. Resting heart rate < 50 or > 100 beats per minute at Screening
23. Oral temperature > / = 38 degrees Celsius (100.4 degrees Fahrenheit)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
The occurrence of AEs | From Day 1 through Day 57
The occurrence of changes in absolute neutrophil count | From Day -1 through Day 91
The occurrence of changes in alanine transaminase (ALT) level | From Day -1 through Day 91
The occurrence of changes in aldolase level | From Day -1 through Day 91
The occurrence of changes in alkaline phosphatase level | From Day -1 through Day 91
The occurrence of changes in aspartate transaminase (AST) level | From Day -1 through Day 91
The occurrence of changes in blood urea nitrogen (BUN) level | From Day -1 through Day 91
The occurrence of changes in calcium level | From Day -1 through Day 91
The occurrence of changes in Complete Blood Count (CBC) with differential | From Day -1 through Day 91
The occurrence of changes in diastolic blood pressure in arm A | From Day -1 through Day 91
The occurrence of changes in diastolic blood pressure in arms B and C | From Day -1 through Day 121
The occurrence of changes in direct bilirubin level | From Day -1 through Day 91
The occurrence of changes in heart rate in arm A | From Day -1 through Day 91
The occurrence of changes in heart rate in arms B and C | From Day -1 through Day 121
The occurrence of changes in hemoglobin level | From Day -1 through Day 91
The occurrence of changes in indirect bilirubin level | From Day -1 through Day 91
The occurrence of changes in oral temperature in arm A | From Day -1 through Day 91
The occurrence of changes in oral temperature in arms B and C | From Day -1 through Day 121
The occurrence of changes in physical examination in arm A | From Day -1 through Day 91
The occurrence of changes in physical examination in arms B and C | From Day -1 through Day 121
The occurrence of changes in platelet count | From Day -1 through Day 91
The occurrence of changes in potassium level | From Day -1 through Day 91
The occurrence of changes in prothrombin time/international normalized ratio (INR) | From Day -1 through Day 91
The occurrence of changes in serum creatinine level | From Day -1 through Day 91
The occurrence of changes in sodium level | From Day -1 through Day 91
The occurrence of changes in systolic blood pressure in arm A | From Day -1 through Day 91
The occurrence of changes in systolic blood pressure in arms B and C | From Day -1 through Day 121
The occurrence of changes in total bilirubin level | From Day -1 through Day 91
The occurrence of changes in total creatine kinase (CK) level | From Day -1 through Day 91
The occurrence of changes in White Blood Cell (WBC) count | From Day -1 through Day 91
The occurrence of clinically significant ECG abnormalities | From Day -28 through Day 1
The occurrence of QT interval abnormalities | From Day -28 through Day 1
The occurrence of SAEs in arm A | From Day 1 through Day 91
The occurrence of SAEs in arms B and C | From Day 1 through Day 121
The presence of protein, blood, or glucose in urine | From Day -1 through Day 91

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time 0 up to the last observed concentration at time t (AUC0-t) for XE02 in arm A | From Day 1 through Day 91
Area under the plasma concentration-time curve (AUC) from time 0 up to the last observed concentration at time t (AUC0-t) for XE02 in arms B and C | From Day 1 through Day 121
Area under the plasma concentration-time curve (AUC) from time 0 up to the last observed concentration at time t (AUC0-t) for XE06 in arm A | From Day 1 through Day 91
Area under the plasma concentration-time curve (AUC) from time 0 up to the last observed concentration at time t (AUC0-t) for XE06 in arms B and C | From Day 1 through Day 121
Area under the plasma concentration-time curve (AUC) from time 0 up to the last observed concentration at time t (AUC0-t) for XE17 in arm A | From Day 1 through Day 91
Area under the plasma concentration-time curve (AUC) from time 0 up to the last observed concentration at time t (AUC0-t) for XE17 in arms B and C | From Day 1 through Day 121
Maximum observed plasma concentration (Cmax) for XE02 in arm A | From Day 1 through Day 91
Maximum observed plasma concentration (Cmax) for XE02 in arms B and C | From Day 1 through Day 121
Maximum observed plasma concentration (Cmax) for XE06 in arm A | From Day 1 through Day 91
Maximum observed plasma concentration (Cmax) for XE06 in arms B and C | From Day 1 through Day 121
Maximum observed plasma concentration (Cmax) for XE17 in arm A | From Day 1 through Day 91
Maximum observed plasma concentration (Cmax) for XE17 in arms B and C | From Day 1 through Day 121
The presence of human anti-human antibodies (HAHA) | Day 1
The presence of human anti-human antibodies (HAHA) | Day 29
The presence of human anti-human antibodies (HAHA) | Day 57
The presence of human anti-human antibodies (HAHA) | Day 91
The presence of human anti-human antibodies (HAHA) for Arms B and C | Day 121
Time to maximum observed plasma concentration (Tmax) for XE02 in arm A | From Day 1 through Day 91
Time to maximum observed plasma concentration (Tmax) for XE02 in arms B and C | From Day 1 through Day 121
Time to maximum observed plasma concentration (Tmax) for XE06 in arm A | From Day 1 through Day 91
Time to maximum observed plasma concentration (Tmax) for XE06 in arms B and C | From Day 1 through Day 121
Time to maximum observed plasma concentration (Tmax) for XE17 in arm A | From Day 1 through Day 91
Time to maximum observed plasma concentration (Tmax) for XE17 in arms B and C | From Day 1 through Day 121

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina, United States